CLINICAL TRIAL: NCT07239245
Title: Efficacy and Safety of Transarterial Chemoembolization (TACE) Combined With Atezolizumab Plus Bevacizumab in Neoadjuvant Therapy for Patients With Hepatocellular Carcinoma: an Open-label, Single-arm, Multicenter, Prospective, Phase II Clinical Study
Brief Title: Study to Evaluate the Efficacy and Safety of Neo-Adjuvant TACE and Atezolizumab Plus Bevacizumab Therapy for High-Risk Recurrent Hepatocellular Carcinamo
Acronym: ATTACH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xinyu Bi, Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5353
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Resectable Hepatocellular Carcinoma With High Risk of Recurrence
Keywords: Hepatocellular Carcinoma; Neoadjuvant therapy; TACE; Atezolizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Bevacizumab + TACE (Experimental): Participants will receive Atezolizumab plus Bevacizumab on Day 1 of a 21-Day cycle, total 5 cycles( Atezolizumab plus Bevacizumab were used in combination for 4 cycles, and Bevacizumab was discontinued in cycle 5. ), after perform 2-3 transarterial chemoembolization procedure on-demand.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Procedure: Transarterial chemoembolization (TACE)

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by IV infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle.
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at a fixed dose of 15 mg/kg on Day 1 of each 21-day Cycle.
Procedure: Transarterial chemoembolization (TACE) — TACE will be performed by clinical demand.

SUMMARY:
This is an open-label, single-arm, multicenter, prospective, phase II clinical study to evaluate the efficacy and safety of TACE combined with Atezolizumab and Bevacizumab as neoadjuvant treatment in Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form available
2. Patients ≥ 18 years and ≤75years of age at time of signing Informed Consent Form
3. Diagnosis of HCC confirmed by histology
4. Initially resectable with high-risk recurrence factors. High-risk features for resected patients include tumor size >5 cm, tumor number >3, vascular invasion (microvascular invasion or macrovascular invasion - Vp1/Vp2 - of the portal vein) and poor tumor differentiation (defined as Grade 3 or 4).

   Up to three tumors, with largest tumor >5 cm regardless of vascular invasion (microvascular invasion or macrovascular invasion of Vp1/Vp2) or poor tumor differentiation (Grade 3 or 4) Four or more tumors, with largest tumor ≤5 cm regardless of vascular invasion (microvascular invasion or macrovascular invasion of Vp1/Vp2) or poor tumor differentiation (Grade 3 or 4) Up to three tumors, with largest tumor ≤5 cm with vascular invasion (microvascular invasion or macrovascular invasion of Vp1/Vp2) and/or poor tumor differentiation (Grade 3 or 4)
5. Measurable disease (at least one target lesion) according to RECIST v1.1 as determined by the investigator
6. Child-Pugh A
7. ECOG PS 0～1
8. No prior locoregional or systemic treatment for HCC
9. Negative HIV test at screening

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma, recurrent HCC and diffuse HCC
2. Clinically diagnosed hepatic encephalopathy in the last 6 months
3. Autoimmune hepatitis (requiring liver puncture)
4. History of organ transplantation
5. Clinical symptoms of pleural effusion, ascites, pericardial effusion, and any history of kidney disease or nephrotic syndrome
6. Treatment with investigational therapy within 28 days prior to initiation of study treatment
7. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or that are at high risk for bleeding
8. A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
9. Known severe allergic reaction to contrast (e.g., anaphylaxis).
10. Pregnancy or lactating women.
11. Inability to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-11-10 (Estimated); Study Completion 2030-11-10 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | At the time of surgery
  pCR rate is defined as the proportion of participants with an absence of residual tumor at the time of surgery, as assessed by central pathological review.

SECONDARY OUTCOMES:
Major Pathologic Response (MPR) Rate | At the time of surgery
  MPR rate is defined as the proportion of participants with =<30% residual viable tumor in the tumor bed at the time of surgery, as assessed by central pathological review.
Relapse-Free Survival (RFS) | Surgery to the first documented recurrence of disease (up to approximately 2 years)
  RFS is defined as the time from surgery to the first documented recurrence of disease (intrahepatic or extrahepatic) according to EASL and/or RECIST v1.1, or death from any cause.
Event-Free Survival (EFS) | Enrollment up to approximately 2 years
  EFS is defined as the time from enrollment to any of the following events (whichever occurs first): disease progression that precludes surgery, as assessed by the investigator according RECIST v1.1; local regional, or distant disease recurrence as measured by EASL and/or RECIST v1.1; or death from any cause.
Overall Survival (OS) | Enrollment to death from any cause (up to approximately 5 years)
  OS is defined as the time from enrollment to death from any cause.
Treatment-related and -unrelated toxicities (AEs, SAEs) according to NCI CTCAE v5.0 | From the start of treatment to 30 days after surgery
  Summary of adverse events by treatment arm and CTCAE (version 5.0) grade and frequency of clinically significant abnormal laboratory parameters.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shanxi Cancer Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No